CLINICAL TRIAL: NCT01117571
Title: A Prospective, Multi-Center Study to Evaluate the ConforMIS iUni® G2 Unicompartmental Knee Resurfacing Device
Brief Title: Multi-Center Study to Evaluate the ConforMIS iUni Knee Implant
Acronym: iUni
Status: Terminated | Type: Observational
Why Stopped: Decision of investigational team
Sponsor: Restor3D (Industry)
Responsible Party: Sponsor
Other Study IDs: 09-001
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis
Keywords: knee; osteoarthritis; unicompartmental; arthroplasty; knee resurfacing; Conformis; patient specific
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- open label: iUni® Unicompartmental Knee Resurfacing Device
  Interventions: Device: iUni® Unicompartmental Knee Resurfacing Device

INTERVENTIONS:
Device: iUni® Unicompartmental Knee Resurfacing Device — The iUni® Unicompartmental Resurfacing Device is an FDA cleared and CE Marked implant designed for patients with damage isolated to either the medial or lateral tibiofemoral compartment of the knee. The patient-specific iUni is designed from a CT scan of an individual patient's knee using a design process which interactively maps the diseased area and defines the extent of misalignment present in the knee. This process allows definition of the shape and size of the femoral and tibial components of the implant, as well as the disposable instrumentation

SUMMARY:
Study is prospective and multi-center. Study will include 100 to 200 patients across up to 20 sites.The study sites will be located in the United States.The study objective is to evaluate the safety and performance of the ConforMIS iUni® Unicompartmental Knee Resurfacing Device in patients with single compartment osteoarthritis.

DETAILED DESCRIPTION:
The iUni G2 Unicompartmental Resurfacing Device (iUni) is an FDA cleared and CE Marked implant designed for patients with damage isolated to either the medial or lateral tibiofemoral compartment of the knee. The study subjects will be followed for 10 years post implant. The study objective is to evaluate the safety and performance of the ConforMIS iUni® Unicompartmental Knee Resurfacing Device in patients with single compartment osteoarthritis. The iUni is a patient-specific unicompartmental resurfacing device designed from the patient's unique anatomy using proprietary software which interprets data from the patient's CT scan. The patient matched implant design is then coupled with unique patient-matched disposable instrumentation designed using the same CT data and software. The follow-up visit schedule will include visits at 6 weeks, 6 months (optional), 1 year, 2 years, 5 years and 10 years post implant.The remaining follow-up data collected at years 3, 4, 6, 7, 8, and 9 may be collected via phone call/email and does not require a subject visit to the site.The study sites will be located in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical condition included in the approved Indications For Use
2. Unicompartmental osteoarthritis of the medial or lateral tibiofemoral compartment
3. Willingness to participate in the clinical study, to give informed consent and to attend all follow-up visits
4. > 18 years of age

Exclusion Criteria:

1. Simultaneous bilateral procedure required
2. BMI > 35
3. Treatment for cancer within the past 5 years, with the exception of skin cancer
4. Poorly controlled diabetes
5. Neuromuscular conditions which prevent patient from participating in study activities
6. Active local or systemic infection
7. Immunocompromised
8. Fibromyalgia or other general body pain related condition
9. Advanced tricompartmental osteoarthritis
10. Symptomatic patellofemoral disease
11. Rheumatoid arthritis or other forms of inflammatory joint disease
12. Loss of bone or musculature, osteoporosis, osteonecrosis, neuromuscular or vascular compromise in the area of the joint to be operated to an extent that the procedure is unjustified
13. Advanced loss of osteochondral structure on the affected femoral condyle
14. Compromised ACL, PCL or collateral ligament
15. Severe (>15º) fixed valgus or varus deformity
16. Extension deficit > 15 º
17. Prior history of failed implant surgery of the joint to be treated
18. Unwilling or unable to comply with study requirements
19. Participation in another clinical study which would confound results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 who have uni-compartmental osteoarthritis to be treated with a unilateral knee resurfacing procedure
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2014-10-30 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Knee Society Score | 2 years
  to assess knee pain and function
WOMAC Osteoarthritis Index | 2 years
  to assess knee pain and function

SECONDARY OUTCOMES:
Knee Society Score and WOMAC at years 5 and 10 post-implantation | 10 years
  Patient reported outcomes measuring pain and function
Annual revision rates at years 1 through 10 post-implantation | 10 years
  Number of revision rates
Incidence of major procedure-related and device-related complications | 10 years
  rate of incidence of serious adverse events that are related to the device or the procedure
Length of tourniquet time in minutes | 6 weeks
  how long the tourniquet was on the patient in surgery
Length of hospital stay in hours | 6 weeks
  How long each patient was in the hospitals from admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: C. Lowry Barnes, M.D, Principal Investigator — Hip Knee Arkansas Foundation; Marc Quartulli, Study Director — Restor3D
Locations (8):
- United States (8):
  - Arkansas Specialty Orthopaedics & HipKneeArkansas Foundation for the Facility, Little Rock, Arkansas
  - S.T.A.R. Orthopaedics, La Quinta, California
  - Center for the Knee and Shoulder, Monterey, California
  - JFK Medical Center, Atlantis, Florida
  - Heekin Clinic, Jacksonville, Florida
  - Great Lakes Bone and Joint, Battle Creek, Michigan
  - Orthopedic Associates of Pittsburgh, Monroeville, Pennsylvania
  - Advanced Orthopedics and Sports Medicine, Cypress, Texas

IPD SHARING:
Plan to Share IPD: No